CLINICAL TRIAL: NCT03609177
Title: Improving Advance Care Planning in Oncology: A Pragmatic, Cluster-Randomized Trial Integrating Patient Videos and Clinician Communication Training
Brief Title: Advance Care Planning: Promoting Effective and Aligned Communication in the Elderly
Acronym: ACP-PEACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Boston Medical Center (Other); Northwell Health (Other); Mayo Clinic (Other); Duke University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, James A. Tulsky, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-276; UG3AG060626 (NIH)
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Other Cancer
Keywords: Cancer Care
MeSH Terms: interventions — Advance Care Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Advance Care Planning (Experimental): -Survey:
  * A group of older patients with advanced cancer (N=450) will have a survey over the course of the 36 months of recruitment.
  * Participants will be provided written copies of the questions to follow along during the interviews
  Interventions: Other: Clinician Communication Skills Training; Other: Advance Care Planning (ACP) Decisions Videos Decisions Aids
- Advance Care Planning-Video Declaration (Experimental): Video Declaration:
  * From among this group of 450 participants, the video declaration of preferences activity will be conducted with 240 patients.
  * For those participants that agree to the video declaration, they will proceed with recording of their video declarations
  * The RA will begin by reading a standardized introduction to aid the subject do the video
  Interventions: Other: Clinician Communication Skills Training; Other: Advance Care Planning (ACP) Decisions Videos Decisions Aids; Other: Video Declarations (ViDec)
- Comprehensive Record Review of ACP (Other): * A review of Medical orders for resuscitation preferences in the electronic health record
  * A review of Medical orders for Palliative care consultations preferences in the electronic health record
  * A review of Medical orders for Hospice use preferences in the electronic health record
  Interventions: Other: Clinician Communication Skills Training; Other: Advance Care Planning (ACP) Decisions Videos Decisions Aids; Other: Video Declarations (ViDec)
- Main Study Arm (Experimental): Patients with cancer being seen at the 30 oncology clinics will be exposed to clinicians who have had communication skills training (Vital Talk) and who are using video decision aids (ACP Decisions). Our main outcome is advance care planning documentation.
  Interventions: Other: Clinician Communication Skills Training; Other: Advance Care Planning (ACP) Decisions Videos Decisions Aids; Other: Video Declarations (ViDec)

INTERVENTIONS:
Other: Clinician Communication Skills Training — Communication skills training
  Other Names: Vital Talk Communication Skills Training
Other: Advance Care Planning (ACP) Decisions Videos Decisions Aids — ACP Decisions video decision aids
Other: Video Declarations (ViDec) — Recording of patient advance care planning videos
  Arms: Advance Care Planning-Video Declaration; Comprehensive Record Review of ACP; Main Study Arm

SUMMARY:
In this research study, the investigators are working to help oncologists better serve patients by delivering more patient-centered, goal-concordant care that may improve health care delivery.

- It is expected that about 30,000 people will take part in this research study, 29,550 of these patients, the vast majority, will be included only for medical record review.

DETAILED DESCRIPTION:
The purpose of this study is to improve the quality of care provided to millions of older Americans with cancer. The investigators are working to help oncologists better serve patients by delivering more patient-centered, goal-concordant care that may dramatically improve health care delivery.

This is pragmatic stepped wedge cluster randomized trial (SW-CRT) of a Comprehensive ACP (Advance Care Planning) Program among older oncology patients. The ACP Program will include training clinicians in communication skills and using video decision aids for participants.

- This study will involve medical record review of 30,000 people age 65 or older with advanced cancer.

We will also recruit 450 eligible patients (150 patients from each of our three sites broken down into 75 patients during the control phase and 75 patients during the intervention phase) to conduct a survey for our secondary patient-centered outcomes (confidence, satisfaction with physician communication, patient decisional satisfaction and regret). From among this sub-group we will engage 240 participants (80 from each of our three sites broken down into 40 patients during the control phase and 40 patients during the intervention phase) in an activity to film video declarations of their preferences.

During the first year, three pilot sites (one at each health care system) will trial the intervention. The subjects recruited at these pilot sites will not be included in the final analysis. Thus, the main trial will begin during year 2 and continue through year 5 with recruitment of 30,000 subjects for the primary outcome at 30 oncology clinics. The first year pilot will serve to inform the larger roll-out and the intervention may change during the first year based on pilot-clinic experience.

ELIGIBILITY:
Inclusion Criteria for clinics:

Clinic eligibility criteria include:

* More than one oncologist
* Serve a patient population that is at least 30% aged 65 or older
* Disease-based oncology clinic

Subject Eligibility: (for the in-person surveys):

- Any patient affiliated with one of the study clinics who speaks English and is aged 65 or older with advanced cancer is eligible for participation. Advanced cancer is defined as metastatic disease for solid tumors and recurrent or refractory disease for hematological malignancies. There are no exclusions based on gender, race, or ethnicity.

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 13800 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A. Tulsky, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Northwell Health, New Hyde Park, New York
  - Duke Health, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Volandes AE, Chang Y, Lakin JR, Paasche-Orlow MK, Lindvall C, Zupanc SN, Martins-Welch D, Carney MT, Burns EA, Itty J, Emmert-Tangredi K, Martin NJ, Sanghani S, Tilburt J, Pollak KI, Davis AD, Garde C, Barry MJ, El-Jawahri A, Quintiliani L, Sciacca K, Goldman J, Tulsky JA. An Intervention to Increase Advance Care Planning Among Older Adults With Advanced Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e259150. doi: 10.1001/jamanetworkopen.2025.9150. PMID 40343696
- [Derived] Lakin JR, Gundersen DA, Lindvall C, Paasche-Orlow MK, Tulsky JA, Brannen EN, Pollak KI, Kennedy D, McLeggon JA, Stout JJ, Volandes A; ACP-PEACE Investigators. A Yet Unrealized Promise: Structured Advance Care Planning Elements in the Electronic Health Record. J Palliat Med. 2021 Aug;24(8):1221-1225. doi: 10.1089/jpm.2020.0774. Epub 2021 Apr 7. PMID 33826860
- [Derived] Lakin JR, Brannen EN, Tulsky JA, Paasche-Orlow MK, Lindvall C, Chang Y, Gundersen DA, El-Jawahri A, Volandes A; ACP-PEACE Investigators. Advance Care Planning: Promoting Effective and Aligned Communication in the Elderly (ACP-PEACE): the study protocol for a pragmatic stepped-wedge trial of older patients with cancer. BMJ Open. 2020 Jul 14;10(7):e040999. doi: 10.1136/bmjopen-2020-040999. PMID 32665394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from April, 2020 - November, 2022. Locations: 36 cancer clinics
Pre-assignment Details: This is a stepped-wedge, cluster randomized trial where clinics were randomized at various steps to move from a control period to the intervention periods. A total of 13,800 unique participants from 29 clinics were enrolled in the study. Participants could have contributed data multiple times during any step of the study.
Units Other Than Participants: clinic
Groups:
- Sequence 1: Control (6 Months), Intervention (24 Months): Clinics participated in a baseline control period for 6 months followed by 24 months of intervention
- Sequence 2: Control (12 Months), Intervention (18 Months): Clinics participated in control periods for 12 months followed by 18 months of intervention
- Sequence 3: Control (18 Months), Intervention (12 Months): Clinics participated in control periods for 18 months followed by 12 months of intervention
- Sequence 4: Control (24 Months), Intervention (6 Months): Clinics participated in control periods for 24 months followed by 6 months of intervention
Period: Baseline
Arm/Group | Sequence 1: Control (6 Months), Intervention (24 Months) | Sequence 2: Control (12 Months), Intervention (18 Months) | Sequence 3: Control (18 Months), Intervention (12 Months) | Sequence 4: Control (24 Months), Intervention (6 Months)
Started | 1571; 6 clinic | 1604; 9 clinic | 1151; 9 clinic | 1376; 5 clinic
Intervention | 0; 0 clinic | 0; 0 clinic | 0; 0 clinic | 0; 0 clinic
Control | 1571; 6 clinic | 1604; 9 clinic | 1151; 9 clinic | 1376; 5 clinic
Completed | 1571; 6 clinic | 1604; 0 clinic | 1151; 0 clinic | 1376; 5 clinic
Not Completed | 0; 0 clinic | 0; 9 clinic | 0; 9 clinic | 0; 0 clinic
Period: Step 1
Arm/Group | Sequence 1: Control (6 Months), Intervention (24 Months) | Sequence 2: Control (12 Months), Intervention (18 Months) | Sequence 3: Control (18 Months), Intervention (12 Months) | Sequence 4: Control (24 Months), Intervention (6 Months)
Started | 1593; 6 clinic | 1538; 9 clinic | 1152; 9 clinic | 1253; 5 clinic
Intervention | 1593; 6 clinic | 0; 0 clinic | 0; 0 clinic | 0; 0 clinic
Control | 0; 0 clinic | 1538; 9 clinic | 1152; 9 clinic | 1253; 5 clinic
Completed | 1593; 6 clinic | 1538; 9 clinic | 1152; 9 clinic | 1253; 5 clinic
Not Completed | 0; 0 clinic | 0; 0 clinic | 0; 0 clinic | 0; 0 clinic
Period: Step 2
Arm/Group | Sequence 1: Control (6 Months), Intervention (24 Months) | Sequence 2: Control (12 Months), Intervention (18 Months) | Sequence 3: Control (18 Months), Intervention (12 Months) | Sequence 4: Control (24 Months), Intervention (6 Months)
Started | 1741; 6 clinic | 1589; 9 clinic | 1033; 6 clinic | 1440; 5 clinic
Intervention | 1741; 6 clinic | 1589; 9 clinic | 0; 0 clinic | 0; 0 clinic
Control | 0; 0 clinic | 0; 0 clinic | 1033; 6 clinic | 1440; 5 clinic
Completed | 1741; 6 clinic | 1589; 9 clinic | 1033; 6 clinic | 1440; 5 clinic
Not Completed | 0; 0 clinic | 0; 0 clinic | 0; 0 clinic | 0; 0 clinic
Period: Step 3
Arm/Group | Sequence 1: Control (6 Months), Intervention (24 Months) | Sequence 2: Control (12 Months), Intervention (18 Months) | Sequence 3: Control (18 Months), Intervention (12 Months) | Sequence 4: Control (24 Months), Intervention (6 Months)
Started | 1961; 6 clinic | 1464; 9 clinic | 1177; 9 clinic | 1485; 5 clinic
Intervention | 1961; 6 clinic | 1464; 9 clinic | 1177; 9 clinic | 0; 0 clinic
Control | 0; 0 clinic | 0; 0 clinic | 0; 0 clinic | 1485; 5 clinic
Completed | 1961; 6 clinic | 1461; 9 clinic | 1177; 9 clinic | 1485; 5 clinic
Not Completed | 0; 0 clinic | 3; 0 clinic | 0; 0 clinic | 0; 0 clinic
Period: Step 4
Arm/Group | Sequence 1: Control (6 Months), Intervention (24 Months) | Sequence 2: Control (12 Months), Intervention (18 Months) | Sequence 3: Control (18 Months), Intervention (12 Months) | Sequence 4: Control (24 Months), Intervention (6 Months)
Started | 1789; 6 clinic | 1519; 9 clinic | 1318; 9 clinic | 1603; 5 clinic
Intervention | 1789; 6 clinic | 1519; 9 clinic | 1318; 9 clinic | 1603; 5 clinic
Control | 0; 0 clinic | 0; 0 clinic | 0; 0 clinic | 0; 0 clinic
Completed | 1789; 6 clinic | 1519; 9 clinic | 1318; 9 clinic | 1603; 5 clinic
Not Completed | 0; 0 clinic | 0; 0 clinic | 0; 0 clinic | 0; 0 clinic

BASELINE CHARACTERISTICS:
Population: No difference
Groups:
- Intervention Arm: Patients with cancer being seen at the 30 oncology clinics will be exposed to clinicians who have had communication skills training (Vital Talk) and who are using video decision aids (ACP Decisions). Our main outcome is advance care planning documentation.
  Clinician Communication Skills Training: Communication skills training
  Advance Care Planning (ACP) Decisions Videos Decisions Aids: ACP Decisions video decision aids
  Video Declarations (ViDec): Recording of patient advance care planning videos
- Usual Care Arm: Patients who were not exposed to any intervention
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Usual Care Arm | Total
Number analyzed (Participants) | 15754 | 13603 | 29357
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.4 (6.6) | 74.6 (6.7) | 74.5 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7284 | 6729 | 14013
  Male | 8470 | 6874 | 15344
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 454 | 392 | 846
  Not Hispanic or Latino | 14750 | 12,801 | 27551
  Unknown or Not Reported | 550 | 410 | 960
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 35 | 27 | 62
  Asian | 556 | 479 | 1035
  Native Hawaiian or Other Pacific Islander | 7 | 3 | 10
  Black or African American | 1978 | 1455 | 3433
  White | 11830 | 10441 | 22271
  More than one race | 1 | 10 | 11
  Unknown or Not Reported | 1347 | 1188 | 2535
Language [Count of Participants; unit: Participants]
  English | 15096 | 13067 | 28163
  Other | 554 | 490 | 1044
  Unknown | 104 | 46 | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Advance Care Planning Documentation
Description: Any advance directive (e.g., living will, POLST, etc.) and changes of resuscitation orders or any indication in the EHR of a goals-of-care or advance care planning conversation
Time Frame: 6 months
Population: The primary outcome measure was assessed at the participant level (all eligible patients) and not at the unit level.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 15754 | 13603
Participants
  Baseline | 0 | 1163
  Step 1 | 349 | 901
  Step 2 | 886 | 511
  Step 3 | 1047 | 259
  Step 4 | 1698 | 0
Statistical Analysis 1: Comparison: Intervention Arm vs Usual Care Arm; Test type: Superiority; p < 0.05, binomial regression with identity link; Risk Difference (RD) = 6.8, 95% CI 2-sided [2.8 to 10.8]

2. Secondary Outcome: Number of Participants With CODE Status Limitations
Description: Documented choices regarding CPR and mechanical ventilation in the EHR
Time Frame: 6 months
Population: The secondary outcome measure was assessed at the participant level (all eligible patients) and not at the unit level.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Arm: Patient Physician Experienced Training
- Usual Care: Usual Care Group
Arm/Group | Intervention Arm | Usual Care
Number analyzed (Participants) | 15754 | 13603
Participants
  Baseline | 0 | 303
  Step 1 | 58 | 205
  Step 2 | 155 | 142
  Step 3 | 280 | 74
  Step 4 | 354 | 0
Statistical Analysis 1: Comparison: Intervention Arm vs Usual Care; Test type: Superiority; p < 0.05, binomial regression with identity link; Risk Difference (RD) = -0.1, 95% CI 2-sided [-0.7 to 0.6]

3. Secondary Outcome: Rate of Palliative Care Consultation
Description: Use of palliative care services (consults, outpatient visits) in the EHR
Time Frame: 6 months
Population: The secondary outcome measure was assessed at the participant level (all eligible patients) and not at the unit level.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 15754 | 13603
Participants
  Baseline | 0 | 531
  Step 1 | 102 | 375
  Step 2 | 324 | 253
  Step 3 | 443 | 128
  Step 4 | 648 | 0
Statistical Analysis 1: Comparison: Intervention Arm vs Usual Care Arm; Test type: Superiority; p < 0.05, binomial regression with identity link; Risk Difference (RD) = 0.7, 95% CI 2-sided [-0.5 to 1.90]

4. Secondary Outcome: Rate of Hospice Use
Description: Use of hospice documented in the EHR
Time Frame: 6 months
Population: The secondary outcome measure was assessed at the participant level (all eligible patients) and not at the unit level.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Patient Physician Experienced Training
- Usual Care: Usual Care
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 15754 | 13603
Participants
  Baseline | 0 | 491
  Step 1 | 50 | 348
  Step 2 | 260 | 202
  Step 3 | 350 | 108
  Step 4 | 468 | 0
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p < 0.05, binomial regression with identity link; Risk Difference (RD) = 0.3, 95% CI 2-sided [-0.4 to 1.0]

5. Secondary Outcome: Confidence in Future Care
Description: (in person survey) patient confidence that they will receive the right care at the right time by their health system. The scale ranged from 1 Not at all confident to 5 Very confident. Higher values represent a better outcome.
Time Frame: 6 months
Population: The secondary outcome measure was assessed at the participant level (all eligible patients) and not at the unit level.
Measure: Count of Participants; unit: Participants
Groups:
- Control: Participants who have filled out a survey from the control group
- Intervention: Participants who have filled out a survey from the intervention group
Arm/Group | Control | Intervention
Number analyzed (Participants) | 196 | 122
Participants
  None to little confidence | 4 | 4
  Somewhat confident | 13 | 8
  Fairly confident | 27 | 15
  Very Confident | 137 | 90
  Unknown | 15 | 5

6. Secondary Outcome: Communication and Decisional Satisfaction
Description: (In person survey) patient satisfaction with communication and decision making.The scale range is from 1- Strongly Disagree to 5 - Strongly Disagree. Higher values represent better outcomes. Subscales were combined questions were summed to compute a total score. The lowest possible score is a 9 and the highest possible score is 45. Lower scores indicate lower communication and decisional satisfaction.
Time Frame: 6 months
Population: The secondary outcome measure was assessed at the participant level (all eligible patients) and not at the unit level.
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 196 | 122
units on a scale | 44 [39 to 45] | 44 [37 to 45]

7. Secondary Outcome: Decisional Regret
Description: (In person survey) patient regret regarding decision making. The response range is 1 - Strongly Disagree to 5 - Strongly agree. Higher numbers represent a worse outcome. Scale questions were summed to compute a total score. The lowest possible score is 2 and the highest possible score is 10. Lower scores indicate less decisional regret.
Time Frame: 6 months
Population: The secondary outcome measure was assessed at the participant level (all eligible patients) and not at the unit level.
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 196 | 122
units on a scale | 2 [2 to 4] | 2 [2 to 4]

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events from baseline up to 4 years and 5.5 months.
Groups:
- Advance Care Planning: -Survey:
  * A group of older patients with advanced cancer (N=450) will have a survey over the course of the 36 months of recruitment.
  * Participants will be provided written copies of the questions to follow along during the interviews
  Clinician Communication Skills Training: Communication skills training
  Advance Care Planning (ACP) Decisions Videos Decisions Aids: ACP Decisions video decision aids
- Advance Care Planning-Video Declaration: Video Declaration:
  * From among this group of 450 participants, the video declaration of preferences activity will be conducted with 240 patients.
  * For those participants that agree to the video declaration, they will proceed with recording of their video declarations
  * The RA will begin by reading a standardized introduction to aid the subject do the video
  Clinician Communication Skills Training: Communication skills training
  Advance Care Planning (ACP) Decisions Videos Decisions Aids: ACP Decisions video decision aids
  Video Declarations (ViDec): Recording of patient advance care planning videos
- Comprehensive Record Review of ACP: * A review of Medical orders for resuscitation preferences in the electronic health record
  * A review of Medical orders for Palliative care consultations preferences in the electronic health record
  * A review of Medical orders for Hospice use preferences in the electronic health record
  Clinician Communication Skills Training: Communication skills training
  Advance Care Planning (ACP) Decisions Videos Decisions Aids: ACP Decisions video decision aids
  Video Declarations (ViDec): Recording of patient advance care planning videos
Arm/Group | Advance Care Planning | Advance Care Planning-Video Declaration | Comprehensive Record Review of ACP | Main Study Arm
All-Cause Mortality (participants affected / at risk) | 0/5702 | 0/5702 | 0/5702 | 3958/5702
Serious Adverse Events (participants affected / at risk) | 0/5702 | 0/5702 | 0/5702 | 0/5702
Other Adverse Events (participants affected / at risk) | 0/5702 | 0/5702 | 0/5702 | 0/5702

LIMITATIONS AND CAVEATS:
Stepped-wedge designs present challenges. Our study occurred entirely during COVID. We assessed ACP documentation in the EHR to measure whether the ix could lead to better communication. We didn't assess the quality of the documentation in the entire sample. We were not able to track video use at the patient level that allowed linkage to either patients or EHR-based outcomes. The video decision aids in this trial are intended to support clinicians who have been trained in communication skills.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT03609177/Prot_SAP_000.pdf